CLINICAL TRIAL: NCT00029445
Title: Evaluation of Viral Factors and Immune Parameters to Study HIV-Specific Immunity
Brief Title: Leukapheresis to Obtain Plasma or Lymphocytes for Studies of HIV-infected Patients, Including Long-term Non-progressors
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 020086; 02-I-0086
Record Dates: First submitted 2002-01-11; First posted 2002-01-14 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-08-28

CONDITIONS: HIV
Keywords: Natural History; Long-term nonprogressors; HLA B*5701; Apheresis; HIV Infection
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Family members: Family members of individuals with innate control over HIV
- HIV infection with one of the following HLA types: B*27+, B*35+,B*44+, B*57+, B*58+, and/or A*02.: People living with HIV with specific HLA-types.
- Long term nonprogressors: Individuals with innate control over HIV

SUMMARY:
This study will collect white blood cells and plasma for research on how the immune system controls HIV infection. The immune system of a very small group of HIV-infected patients, called non-progressors, has been able to control HIV for long periods without antiretroviral therapy. Some immune system-related genes important for this control have been identified in these patients. This study will examine the contribution of HLA genes B*57+, B*27+ and A*01+ to HIV disease in progressors and long-term non-progressors. (HLA type is a genetic marker of the immune system.)

HIV-infected patients 18 years of age and older with HLA types B*57+, B*27+ and/or A*01+ may be eligible for this study.

Participants will undergo apheresis-a method for collecting larger quantities of certain blood components than can safely be collected through a simple blood draw-by one of the following two methods:

* Automated pheresis - Blood is drawn through a needle placed in an arm vein and spun in a machine, separating the blood components. The white cells are extracted and the red cells, with or without plasma (liquid part of the blood), are re-infused into the donor through the same needle or a needle in the other arm. An anticoagulant (medication to prevent blood from clotting) is usually added to the blood while in the machine to prevent it from clotting during processing.
* Manual pheresis - One unit (1 pint) of blood is drawn through a needle placed in an arm vein, similar to donating a pint of whole blood. The red blood cells, with or without plasma, are separated from the rest of the blood and re-infused to the donor through the same needle. Manual pheresis will be done only when a person s estimated total blood volume or red cell count is too low to safely permit removal of blood through a pheresis machine. An adult small in size or markedly anemic, for example, may fall into this category.

Some of the blood collected through apheresis may be stored for future studies of HIV disease and immune function and for HLA testing, a genetic test of markers of the immune system. Some of the blood may be used to screen for different types of viral liver infections, such as hepatitis A, B, C, D, E, F, or G.

...

DETAILED DESCRIPTION:
In an attempt to elucidate the mechanism(s) of immune-mediated restriction of HIV viral replication, we aim to study three groups of individuals:

1. People living with HIV, who appear to control HIV primarily through virus-specific cellular immunity (long-term nonprogressors/LTNP);
2. People living with HIV who have broadly cross-neutralizing antibody activity against HIV; and
3. the family members of participants exhibiting immunologic control of HIV infection. Although most of our previous efforts have focused on investigating the virus-specific immune responses in a unique group of patients termed LTNP who control HIV by cellular immune-mediated mechanisms, more recently, another group of rare individuals who naturally develop broadly cross-neutralizing antibody activity against HIV isolates have also been identified in our laboratory. Passive transfer studies in nonhuman primates have demonstrated that neutralizing antibodies detectable in a subject at the time of challenge can protect from infection. We aim to recruit more of these participants in an effort to further characterize and compare their virus-specific cellular and humoral immune responses with those in individuals experiencing progressive infection. As we attain greater insight into differences between these participant groups, we hope to perform genetic studies that would enable us to more precisely identify susceptibility or protective genes, which could be potentially used to construct a familial pedigree. We anticipate that all of these findings will contribute to an enhanced understanding of the nature of effective HIVspecific humoral and cellular immunity, which will help focus future vaccine design efforts. For our studies, it will be necessary to obtain larger quantities of plasma or mononuclear cells than can be safely obtained by simple phlebotomy. These components can be easily and safely obtained using apheresis procedures in the Clinical Center Apheresis Unit. This protocol is designed to conform to the requirements of the Apheresis Unit for donors to have leukapheresis or plasmapheresis procedures. In select participants, lymphocytes obtained from lymph node biopsy will also be studied.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Adult (18 years-old or older)
  2. Eligibility to undergo apheresis procedures; or, for participants who are unable to undergo apheresis, willingness to undergo blood draw for research purposes that remain within safety guidelines established by NIH policy.
  3. Willingness to give informed consent for the storage of blood or tissue samples and HLA testing

AND at least one of the following:

* An HIV-seropositive participant categorized as an LTNP as defined by clinical and laboratory criteria, regardless of HLA class I type.
* HIV-seropositive progressors
* Persons who are seronegative for HIV but are family members of seropositive participants exhibiting immunologic control of HIV

EXCLUSION CRITERIA:

1. Pregnant
2. Cardiovascular instability, severe anemia, inadequate venous access, severe coagulation disorder, or any other condition that the Principal Investigator or Apheresis Unit staff considers a contraindication to the apheresis procedure or research blood draw.
3. Any condition that, in the opinion of the investigator, contraindicates participation in this study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals identified as having innate control over the HIV virus
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2001-08-09 (Actual)

PRIMARY OUTCOMES:
To further investigate differences in the virus-specific T cell-mediated responses between HIV-1-infected LTNP and patients with progressive disease who bear HLA class I alleles that have been associated with delayed disease progression and to c... | Ongoing
  deeper understanding of the components and correlates of an effective HLA class-I-restricted HIV-specific CD8+ T cell response
Perform genetic studies to characterize immune-related susceptibility/protective genes and compare these between patients groups and within families. | Ongoing
  Availability of cells from family members of LTNP with or without putative response modifiers could help in defining the role of these genes in shaping the immune response to HIV.
Identify patients with broadly neutralizing sera and characterize their HIV-specific B cell responses | Ongoing
  characterize HIV-specific neutralizing antibody activity
Identification of the cause and effect relationships between viremia and putative immune correlates of control of HIV replication | Ongoing
  to understand HIV-specific immunity

CONTACTS AND LOCATIONS:
Overall Officials: Daniel C Rogan, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underline the results reported in the publication, after deidentification (text, tables, figures, and appendices)
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose. Analysis for individual participant data meta-analysis. Proposals may be submitted up to 36 months following article publication.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2002-I-0086.html